CLINICAL TRIAL: NCT00099307
Title: An Exploratory Study on Detection of Cortical Damage in Patients With Multiple Sclerosis Using Magnetic Resonance Imaging
Brief Title: Magnetic Resonance Imaging to Detect Brain Damage in Patients With Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050039; 05-N-0039
Record Dates: First submitted 2004-12-10; First posted 2004-12-10 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-09-28

CONDITIONS: Multiple Sclerosis
Keywords: White Matter; Grey Matter; Brain; Disability; Lesions; Multiple Sclerosis; MS; Healthy Volunteer; HV
MeSH Terms: conditions — Multiple Sclerosis

SUMMARY:
This study will determine whether magnetic resonance imaging (MRI) can detect damage to certain parts of the brain and analyze the thickness of the brain's outer surface in patients with multiple sclerosis. MRI is a diagnostic test that uses a strong magnetic field and radio waves to obtain images of body organs and tissues. It can sometimes permit diagnosis even before symptoms develop.

MS is a disease of white matter, the fatty covering around the nerves in the brain and spinal cord. The nerves themselves are called gray matter. Damage to white matter impairs nerve function, leading to a variety of symptoms, such as weakness, vision problems, difficulty walking, paralysis, and others. MRI can detect some changes in white matter, but changes that may also appear in gray matter may be more difficult to find. This study will use new MRI techniques to try to identify gray matter damage in patients with MS.

Healthy volunteers and people with MS or clinically isolated syndrome (an early stage of MS in which the patient has had just one of the problems MS can cause) who are between 18 and 55 years of age may be eligible for this study. Candidates are screened with a medical history and neurological examination, and blood and urine tests.

Within one month of the screening evaluation, participants undergo MRI scanning on a standard 1.5 Tesla machine to confirm their health status. (The power of the MRI scanner is measured in Tesla; the higher the Tesla, the better the visualization.) For this procedure, the subject lies on a table that moves into the scanner (a narrow cylinder with a magnetic field), and wears earplugs to muffle loud knocking and thumping sounds that occur during the scanning process. During the procedure, a contrast agent called Gadolinium is injected into the blood stream to brighten the images. The test lasts about 2 hours, during which time the subject must lie still for up to a few minutes at a time.

Within a month after the first MRI, participants repeat the test for a second time. The procedure is identical to the first scan, except a 3.0 Tesla machine is used.

DETAILED DESCRIPTION:
OBJECTIVE: Detection of cortical lesions in patients with multiple sclerosis (MS) using magnetic resonance imaging (MRI) is challenging. Their identification might provide more insight in explaining the level of disability in patients with MS.

Primary aim of the present study is identifying cortical lesions in patients with MS using MRI. As a secondary aim, correlation between cortical lesions presence and clinical disability score (i.e. Expanded Disability Status Score or EDSS scale) will be analyzed. Tertiary aims will be provided by the relationships between the presence of cortical lesions and reduction in cortical thickness and extent of remote white matter disease pathology. Additionally, the role of white matter lesions in causing remote pathology will be studied. To better characterize this damage, patients with previous stroke, presenting with a single lesion on the pyramidal tract will be enrolled and diffusion-derived indices of white matter remote tracts will be computed.

STUDY POPULATION: Fifty patients with definite MS or with a single attack and an MRI suggestive of MS (i.e., clinically isolated syndrome) according to McDonald criteria, and 55 healthy volunteers will be enrolled. Fifteen patients with previous ischemic stroke and 15 age- and gender-matched healthy volunteers will also be enrolled.

DESIGN: After a clinical evaluation and an MRI at 1.5 Tesla, each individual will be imaged once at 3.0 Tesla scan. Clinical MRI before and within 15 minutes after contrast injection will be obtained in each patient at both 1.5 and 3 Tesla scans. In addition, 3 spoiled gradient-echo sequence, diffusion tensor images and double inversion recovery sequences will be acquired on the 3 Tesla MRI. Some healthy volunteers (up to 15) and patients (up to 15) will be required to be imaged twice on the 3T magnet as to optimize the sequences of this study. Additionally, 20 patients in whom cortical lesions will be identified using the above-mentioned techniques and 20 healthy volunteers will undergo brain perfusion MRIs. This may represent the third 3T MRI for the former in some instances.

OUTCOME MEASURES: In MS patients, the number of cortical lesions will be computed. The EDSS score will serve for investigating the relationship between cortical lesions and clinical disability. Effect of cortical or white matter lesions in causing remote degeneration will be studied using diffusion tensor and magnetization transfer imaging in patients with both stroke and MS.

ELIGIBILITY:
* INCLUSION CRITERIA - MULTIPLE SCLEROSIS PATIENTS:

Diagnosis of clinically isolated syndrome or MS.

Age between 18 and 55.

EDSS between 0 and 6.5.

EXCLUSION CRITERIA - MULTIPLE SCLEROSIS PATIENTS:

Presence of clinical relapse at the time of the enrollment or within the previous 3 months.

Concomitant systemic disorder or central nervous system diseases of any kind or other related risk factors.

Previous history of alcohol and substances abuse.

Medical contraindications for MRI.

Psychological contraindications for MRI.

Pregnancy.

Unable to provide informed consent.

INCLUSION CRITERIA - HEALTHY VOLUNTEERS:

Age greater than 18 years.

EXCLUSION CRITERIA - HEALTHY VOLUNTEERS:

Systemic disorder or central nervous system diseases of any kind or other related risk factors.

Previous history of alcohol and substances abuse.

Medical contraindications for MRI.

Psychological contraindications for MRI.

Pregnancy.

Unable to provide informed consent.

INCLUSION CRITERIA - STROKE PATIENTS:

Age greater than 18 years.

Pure motor hemiparesis secondary to a first and single acute ischemic infarct localized in the white matter of the pyramidal tract (confirmation and location stroke by MRI).

No other major diseases of the central nervous system or neurological signs.

No other visible MRI lesions of the corticospinal tract on T2-weighted images (e.g., patients with white matter lesions on tracts not connected with the pyramidal tract and clinically silent will not be excluded).

EXCLUSION CRITERIA - STROKE PATIENTS:

Stroke onset less than 3 months prior to the study enrollment.

Previous history of alcohol and substances abuse.

Medical contraindications for MRI.

Contraindications for MRI.

Critical stenosis of either carotids or vertebrobasilar artery as demonstrated by a Transcranial Doppler.

Pregnancy.

Unable to provide informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2004-12-08; Study Completion 2011-09-28

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] McFarland HF. The emerging role of MRI in multiple sclerosis and the new diagnostic criteria. Mult Scler. 2002 Feb;8(1):71-2. doi: 10.1177/135245850200800114. No abstract available. PMID 11936491
- [Background] Li DK, Zhao G, Paty DW. T2 hyperintensities: findings and significance. Neuroimaging Clin N Am. 2000 Nov;10(4):717-38 ,ix. PMID 11359721
- [Background] Harris JO, Frank JA, Patronas N, McFarlin DE, McFarland HF. Serial gadolinium-enhanced magnetic resonance imaging scans in patients with early, relapsing-remitting multiple sclerosis: implications for clinical trials and natural history. Ann Neurol. 1991 May;29(5):548-55. doi: 10.1002/ana.410290515. PMID 1859184